CLINICAL TRIAL: NCT05716451
Title: Randomised Pilot Study on Device-assisted Mobilisation With a Sit/Stand Stabiliser of Critically Ill Patients With Ventilatory Support
Brief Title: Pilot Study on Device-assisted Mobilisation of Critically Ill Patients
Acronym: LIANA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIANA-I
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Muscle Weakness; Critical Illness
Keywords: ICUAW; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Mobilization incl. support by the Liana. In the intervention group, Liana is used to train trunk stability in a sitting position. If this is successful, the patient is trained to stand. Mobilization to higher levels is performed according to clinical standards.
  Interventions: Device: Device-assisted mobilisation with the sit/stand stabilizer Liana
- Control Group (No Intervention): Standard of Care without the use of the Liana. In the control group the therapy is carried out according to the ward standard without using the Liana.

INTERVENTIONS:
Device: Device-assisted mobilisation with the sit/stand stabilizer Liana — Non-invasive device-assisted mobilisation with LIANA
  Arms: Intervention Group

SUMMARY:
This Pilot study will hypothesize that patients with organ insufficiency and breathing assistance in our post-anaesthesia care unit (PACU) and ICU will be mobilized more often to an ICU mobility scale (IMS) ≥ 4 (i.e. standing) using the Liana® mobilizer. Therefore a randomized controlled pilot study will be conducted. The aim is to achieve an important physical function mile stone more often using this device.

Secondary hypotheses are:

1. The intervention will relieve the burden of the health care staff in the unit
2. The intervention will positively influence the functional outcome of critically ill patients
3. The intervention is perceived as positive by the patients

DETAILED DESCRIPTION:
Patients who have been treated in the ICU for a prolonged period of time often have a high degree of immobility. In this context, a state of generalized weakness associated with muscle atrophy (ICUAW) develops in approximately 40% of ICU patients. The severity of generalized weakness may be individual in each patient. It is certain that especially elderly patients and patients with prolonged immobilization have an increased incidence of ICUAW. Symptoms can be highly variable depending on the severity of the course. Some patients report weakness of the extremities to paresis and weakness of the respiratory muscles. Weakness of the respiratory musculature can lead to a prolonged weaning process of mechanical ventilation, prolonging the stay in the ICU. Functional impairments due to ICUAW may also persist many years after the ICU stay. If ICUAW is diagnosed promptly, outcome can be improved by targeted early mobilization. Early mobilization is defined as mobilization in the first 72 h from ICU admission. However, there are numerous barriers to the implementation of early mobilization in critically ill patients, so this remains a major challenge.

Various studies have shown that patients can benefit from a high level of mobilization. For example, Scheffenbichler et al. showed that a high dose of mobilization was associated with increased independence of patients after discharge. The level of mobilization showed positive effects not only in this study, but also in Paton and colleagues. They were able to show that achieving a higher level of mobility (according to the Intensive Care Mobility Scale) was associated with improved outcome at six months. They found that achieving a higher level of mobilization positively affected the health status of patients, whereas increasing the number of mobilizations did not.

With device-assisted mobilization, patients could be mobilized to standing position early and more frequently. The aim of this pilot study is to test whether mobilization of critically ill patients with ventilatory support using device-assisted mobilization leads to increased mobilization to standing (IMS 4) or beyond.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patient with ventilatory support and an expected intensive care stay of at least another 48 h
* Age ≥ 18 years
* Current length of intensive care stay < 48 h

Exclusion Criteria:

* Moribund and critically ill
* Suspected 6-month mortality > 75%.
* Increased intracranial pressure
* Critically ill after cardiopulmonary resuscitation
* Critically ill with primary neuromuscular disease or motor neuron disease
* One or more amputated extremities
* Patients, within 2h after surgery
* Unstable fractures
* Severe traumatic brain injury (e.g., brain and skull injuries)
* Circulatory instability with norepinephrine > 0.3 µg/kg/min
* Patients for whom there is an indication for deep sedation (RASS -5)
* Language barrier
* Fitting of legs into leg trays is not possible due to e.g. patient weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Level of mobilisation (IMS) | 28 Days
  Mean level of mobilisation measured with the Intensive Car Unit Mobility Scale (IMS) till ICU discharge (or Day 28); IMS ranges from 0 (no mobilization) to 10 (independent walking)

SECONDARY OUTCOMES:
Frequency of IMS ≥ 4 | 28 Days
  Frequency of Days with IMS ≥ 4 till ICU discharge (or Day 28)
Handgrip strength | 28 Days
  Muscle strength measured using handgrip strength till ICU discharge (or Day 28)
MRC Sum Score | 28 Days
  Muscle strength measured using Medical Research Council (MRC) Sum Score till ICU discharge (or Day 28); MRC Sum Score ranges from 0 to 60, with 0 worst value
Diaphragma function | 28 Days
  Diaphragm function by diaphragmatic thickening fraction using ultrasound till ICU discharge (or Day 28)
CPAx Score | 28 Days
  The Chelsea Critical Care Physical Assessment Tool (CPAx) during the ICU stay (or till Day 28); ranging from 0 to 50 with 0 the worst score
Trunk Control Test | 28 Days
  Trunk stability using the trunk control test during the ICU stay (or till Day 28)
Duration of MV | 180 Days
  Duration of mechanical ventilation (MV) in days
Patient satisfaction with VRS | 28 Days
  Patient satisfaction with mobilisation using a verbal rating scale (VRS 0-10), 0 the worst score
Staff satisfaction with VRS | 28 Days
  Staff satisfaction with mobilisation using a verbal rating scale (VRS 0-10), 0 being worst score
Staff binding time | 28 Days
  Staff binding time for mobilisation during the ICU stay (or Day 28)
ICU LOS | 180 Days
  ICU length of stay in Days
Hospital LOS | 180 Days
  Hospital length of stays
Time in rehabilitation and hospital | 180 Days
  Time in rehabilitation facilities or hospital in days
(I)ADL | 180 Days
  (Intrumental) Activities of Daily Living Score as measured by Iwashyna et al.; range 0-11, 0 the worst
Disability | 180 Days
  Disability measured with the WHODAS 2.0 score
Quality of life | 180 Days
  Quality of life measured with the EQ-5D-5L. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Detail information is available at https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/
Physical Function | 180 Days
  Physical function measured with the Barthel Score, scoring from 0-100 with 0 the worst

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The plan is to share deidentified data by reasonable scientific request and after signing an appropriate agreement.